CLINICAL TRIAL: NCT05727436
Title: The Effect of Oral Probiotics Containing Streptococcus Salivarius M18 on Gingivitis and Oral Hygiene: A Randomized Clinical Trial
Brief Title: The Effect of Probiotics on Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18081213
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-02

CONDITIONS: Gingivitis; Chronic
MeSH Terms: conditions — Gingivitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel Assignment double-blind, randomized, two-arm parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation concealment will be performed by the use of sealed containers numbered by a "third party" (person, who will not participate in the study). The tablets in the bottles without any titles will be placed in the containers. The tablets in different groups will look similar. The patient on enrollment will receive a container with tablets. Each patient will receive a sealed container with tablets on enrollment. Neither patients nor researchers will be aware of the type of a tablets received by each patient (double blinding).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - probiotic (Experimental): Experimental: Group 1 - probiotic The use of Streptococcus salivarius M18 containing tablets ("Dentoblis", registration number: AM.01.06.01.003.R.000061.07.20; 15.07.2020, MEDICO DOMUS, d.d.o.; 18116, Nis, Serbia)) once a day for 4 weeks (before bedtime after evening brushing).
  Ingredients: basic active ingredients - Streptococcus salivarius M18 (≥5×108 CFU in 1 tablet), Vitamin D (320 IU (8 mcg) in 1 tablet); excipients - isomalt (sweetener), magnesium stearate (vegetable), mint flavoring.
  Interventions: Dietary Supplement: Dentoblis
- Group 2 - placebo (Placebo Comparator): The use of placebo tablets once a day for 4 weeks (before bedtime after evening brushing).
  Ingredients: isomalt (sweetener), magnesium stearate (vegetable), mint flavoring.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dentoblis — Dissolve the tablets in the mouth once a day for 4 weeks
  Other Names: Probiotic: Streptococcus salivarius M18
  Arms: Group 1 - probiotic
Dietary Supplement: Placebo — Dissolve the tablets in the mouth once a day for 4 weeks
  Arms: Group 2 - placebo

SUMMARY:
The aim of the study is to assess the effect of oral probiotics containing Streptococcus salivarius M18 on gingivitis and oral hygiene in young adults.

DETAILED DESCRIPTION:
This will be a double-blind, randomized, placebo-controlled two-arm parallel-group study of the effect of oral probiotics containing Streptococcus salivarius M18 on gingivitis and oral hygiene. The groups will include young adults with gingivitis diagnosed clinically. To assess the effect of oral probiotics, the following parameters will be used: gingival index, GI; gingival bleeding index, GBI and oral hygiene level (the Turesky Modification of the Quigley-Hein Plaque Index, TMQHPI).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-25 years
* Permanent bite;
* Presence of more than 20 teeth;
* Absence of systemic and chronic diseases;
* The diagnosis of gingivitis stated clinically.

Exclusion Criteria:

* Presence of mild, moderate or severe chronic periodontitis;
* Refusal to sign informed consent;
* Taking supplements and medication containing probiotics or prebiotics 1 months before the study;
* Taking antibiotics (within 3 months before the study);
* Allergy to the components of the drugs used in the study;
* Presence of immunodeficiency, taking immunosuppressants.
* Use of other hygiene products, immunostimulants and antibacterials, probiotics, prebiotics during the study;
* Refusal to take a given medication;
* Failure to attend check-ups.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of gingival inflammation using Gingival Index (GI) by H. Loe and J. Silness | 4 weeks after the baseline
  GI is used to assess visual symptoms of gingivitis on mesial, distal, vestibular, and oral areas of each scorable tooth (1.6, 1.2, 2.4, 3.6, 3.2, 4.4). Each area is given a score from 0 to 3. Values are presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e., 0-3). Scoring is performed using standard dental light: 0 = absence of inflammation; 1 = mild inflammation - slight change in color and little change in texture; 2 = moderate inflammation - moderate glazing, redness, oedema, and hypertrophy, bleeding on pressure; 3 = severe inflammation - marked redness and hypertrophy, tendency to spontaneous bleeding, ulceration. Lower scores indicate better results.
Evaluation of gingival inflammation using Gingival Index (GI) by H. Loe and J. Silness | 8 weeks after the baseline
  GI is used to assess visual symptoms of gingivitis on mesial, distal, vestibular, and oral areas of each scorable tooth (1.6, 1.2, 2.4, 3.6, 3.2, 4.4). Each area is given a score from 0 to 3. Values are presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e., 0-3). Scoring is performed using standard dental light: 0 = absence of inflammation; 1 = mild inflammation - slight change in color and little change in texture; 2 = moderate inflammation - moderate glazing, redness, oedema, and hypertrophy, bleeding on pressure; 3 = severe inflammation - marked redness and hypertrophy, tendency to spontaneous bleeding, ulceration. Lower scores indicate better results.
Evaluation of gingival inflammation using Gingival bleeding index (GBI) by J. Ainamo and I. Bay, 1975 | 4 weeks after the baseline
  GBI is used to assess bleeding elicited on probing as a measure of gingival condition. Gingivae are air dried and examiner assesses bleeding using a probe which is gently inserted into gingival crevice to depth of app 1 mm and run around tooth (angle of app 60 deg to long axis of tooth), gently stretching epithelium while sweeping from interproximal to interproximal along sulcular epithelium. BI is assessed on mesial, distal, vestibular, and oral areas of each scorable tooth (whole mouth). Values are presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e., 0-1). BI score:0=no bleeding after 10 sec, 1=bleeding upon probing after 10 sec or immediate bleeding. Lower scores indicate better results.
Evaluation of gingival inflammation using Gingival bleeding index (GBI) by J. Ainamo and I. Bay, 1975 | 8 weeks after the baseline
  GBI is used to assess bleeding elicited on probing as a measure of gingival condition. Gingivae are air dried and examiner assesses bleeding using a probe which is gently inserted into gingival crevice to depth of app 1 mm and run around tooth (angle of app 60 deg to long axis of tooth), gently stretching epithelium while sweeping from interproximal to interproximal along sulcular epithelium. BI is assessed on mesial, distal, vestibular, and oral areas of each scorable tooth (whole mouth). Values are presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e., 0-1). BI score:0=no bleeding after 10 sec, 1=bleeding upon probing after 10 sec or immediate bleeding. Lower scores indicate better results.

SECONDARY OUTCOMES:
Evaluation of oral hygiene using Turesky Modification of the Quigley-Hein Plaque Index | 4 weeks after the baseline
  A plaque detection solution is used to detect the presence of plaque on both the vestibular and oral surfaces of all teeth except the third molars. Each surface is divided into 3 segments: mesial, central and distal. Thus, 6 segments are evaluated for each tooth. Evaluation criteria: 0 - no staining;
  1. - separate areas of plaque in the cervical part;
  2. - plaque in the form of a thin continuous band up to 1 mm wide in the cervical part;
  3. - cervical part is covered by plaque that is more than 1 mm wide, but less than 1/3 of the tooth crown;
  4. - plaque covers 1/3 to 2/3 of the crown;
  5. - plaque covers more than 2/3 of the crown.
Evaluation of oral hygiene using Turesky Modification of the Quigley-Hein Plaque Index | 8 weeks after the baseline
  A plaque detection solution is used to detect the presence of plaque on both the vestibular and oral surfaces of all teeth except the third molars. Each surface is divided into 3 segments: mesial, central and distal. Thus, 6 segments are evaluated for each tooth. Evaluation criteria: 0 - no staining;
  1. - separate areas of plaque in the cervical part;
  2. - plaque in the form of a thin continuous band up to 1 mm wide in the cervical part;
  3. - cervical part is covered by plaque that is more than 1 mm wide, but less than 1/3 of the tooth crown;
  4. - plaque covers 1/3 to 2/3 of the crown;
  5. - plaque covers more than 2/3 of the crown.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Dentistry of Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babina K, Salikhova D, Polyakova M, Svitich O, Samoylikov R, Ahmad El-Abed S, Zaytsev A, Novozhilova N. The Effect of Oral Probiotics (Streptococcus Salivarius k12) on the Salivary Level of Secretory Immunoglobulin A, Salivation Rate, and Oral Biofilm: A Pilot Randomized Clinical Trial. Nutrients. 2022 Mar 7;14(5):1124. doi: 10.3390/nu14051124. PMID 35268099
- [Derived] Babina K, Salikhova D, Doroshina V, Makeeva I, Zaytsev A, Uvarichev M, Polyakova M, Novozhilova N. Antigingivitis and Antiplaque Effects of Oral Probiotic Containing the Streptococcus salivarius M18 Strain: A Randomized Clinical Trial. Nutrients. 2023 Sep 6;15(18):3882. doi: 10.3390/nu15183882. PMID 37764667